CLINICAL TRIAL: NCT06015464
Title: An Ambispective Cohort Study of Orelabrutinib in Combination With Standard Treatment Regimen for Untreated DLBCL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-SR-190
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma, Large B-Cell, Diffuse Neoplasms by Histologic Type
MeSH Terms: conditions — Lymphoma | interventions — orelabrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective cohort: To retrospectively collect information on DLBCL patients treated with orelabrutinib in combination with standard first-line regimens, pooled analysis of the association between recent efficacy and patient characteristics (including biomarkers) in different types of patients to assess the predictive value of ctDNA for prognosis and subsequent therapeutic adjustments during treatment
  Interventions: Drug: Orelabrutinib
- Prospective cohort: Prospective observation to collect information on the efficacy of orelabrutinib in combination with standard treatment regimens in specific types of populations (with a focus on genotyped patients such as MCD, BN2 and N1 subtypes) to validate the predictive value of ctDNA in diagnosis and treatment
  Interventions: Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib — Addition of novel BTK inhibitor, Orelabrutinib，150 mg qd, to standard treatment regimens, which include R-CHOP and Pola-R-CHP

SUMMARY:
To retrospectively collect information on DLBCL patients treated with orelabrutinib in combination with standard first-line regimens, pooled analysis of the association between recent efficacy and patient characteristics (including biomarkers) in different types of patients to assess the predictive value of ctDNA for prognosis and subsequent therapeutic adjustments during treatment; Prospective observation to collect information on the efficacy of orelabrutinib in combination with standard treatment regimens in specific types of populations (with a focus on genotyped patients such as MCD, BN2 and N1 subtypes) to validate the predictive value of ctDNA in diagnosis and treatment. Standard treatment regimens include the R-CHOP regimen and the Pola-R-CHOP regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years Diffuse large B-cell lymphoma (DLBCL) diagnosed by histopathology of the tumour, without any previous anti-tumour therapy or after ≤2 cycles of R-CHOP(like) or Pola-R-CHP therapy only
* Have a clear efficacy evaluation
* Patients eligible for Non-GCB or extra-nodal or dual expression or who, in the judgement of the investigator, would benefit from treatment with Orelabrutinib following genetic testing.
* Patients treated with at least 2 cycles of orelabrutinib in combination with an R-CHOP(like) or Pola-R-CHP regimen

Exclusion Criteria:

* Lymphoma involving the central nervous system or soft meningeal metastases
* Transforming lymphoma, i.e. from other types of lymphoma such as follicular lymphoma, marginal zone lymphoma or chronic lymphocytic leukaemia or small B-cell lymphoma
* Primary mediastinal large B-cell lymphoma
* Patients with poorly controlled cardiovascular disease, infectious disease, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Untreated Diffuse large B-cell lymphoma (DLBCL) patients
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
CR rate of EOT | at the end of Cycle 6-8 (each cycle is 28 days)
  CR rate at the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No